CLINICAL TRIAL: NCT03476109
Title: Predictive Factors and Magnitude of Response to Omalizumab and Mepolizumab in Allergic and Eosinophilic Severe Asthma: a Pragmatic Multicenter Trial in Belgium.
Brief Title: Study of Magnitude and Prediction of Response to Omalizumab and Mepolizumab in Adult Severe Asthma.
Acronym: PREDICTUMAB
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: University Hospital, Ghent (Other); University of Liege (Other); CHU de Charleroi (Other); Erasme University Hospital (Other); Centre Hospitalier Universitaire UCLouvain Namur (Other); Universitair Ziekenhuis Brussel (Other); Brugmann University Hospital (Other); Grand Hôpital de Charleroi (Other); AZ Delta (Other); Centre Hospitalier Universitaire Saint Pierre (Other); KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/19JUI/325; PNEU-ASTHMA-02 (Other: CUSL); 2017-002473-19 (EudraCT Number)
Record Dates: First submitted 2017-10-17; First posted 2018-03-23 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Severe Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Severe asthma patients who are eligible to both anti-IgE (omalizumab) and anti-IL-5 (mepolizumab) therapies, will be randomized to decide the first treatment to start. Patients will then be prolonged or switched to the other according to the clinical response. There will be 5 possibilities: oma(lizumab) group, mepo(lizumab) group, oma-mepo switch, mepo-oma switch, and oma/mepo failure.
Who Masked: Outcomes Assessor
Masking Description: The analysis of the response rate and magnitude, as well as of biomakers predicting the response, will be performed by an independent assessor and a biostatistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Omalizumab (Active Comparator): Patients randomized to omalizumab and then prolonged or not (based on their response at 4 months) until the end of the study (22mo).
  Non responders will be switched to mepolizumab arm.
  Interventions: Drug: Randomisation to mepolizumab
- Mepolizumab (Active Comparator): Patients randomized to mepolizumab and then prolonged or not (based on their response at 6 months) until the end of the study (22mo).
  Non responders will be switched to omalizumab arm.
  Interventions: Drug: Randomisation to omalizumab

INTERVENTIONS:
Drug: Randomisation to omalizumab — The only intervention will be that allocation of patients to omalizumab or mepolizumab (to both of which patients will be eligible) will be randomized, to avoid that the initial decision is biased by confounding factors that are likely, but unproven, to affect the treatment response. Then, in case of non-response, patients will be switched to the other drug, as routine clinical practice would indicate.
  Other Names: Active-controlled
  Arms: Mepolizumab
Drug: Randomisation to mepolizumab — The only intervention will be that allocation of patients to omalizumab or mepolizumab (to both of which patients will be eligible) will be randomized, to avoid that the initial decision is biased by confounding factors that are likely, but unproven, to affect the treatment response. Then, in case of non-response, patients will be switched to the other drug, as routine clinical practice would indicate.
  Other Names: Active-controlled
  Arms: Omalizumab

SUMMARY:
Pragmatic trial to define the magnitude and the predictive factors of the response to omalizumab and mepolizumab in adult patients with severe refractory asthma and eligible to both therapies.

DETAILED DESCRIPTION:
Title "PREDICTUMAB: Predictive factors and magnitude of response to omalizumab and mepolizumab in allergic and eosinophilic severe asthma: a multicenter, open, active-controlled, randomized trial in adult patients in Belgium".

Rationale and background New treatments are now available to treat severe refractory asthma, which affects about 3 to 5% of asthma patients. In particular, biological therapies using monoclonal antibodies targeted to immunoglobulin E (IgE) or interleukin (IL)-5 (and in the future other cytokines or growth factors) benefit to certain patients. Identifying those patients who will better benefit from a specific treatment requires the validation of features (clinical traits, biomarkers) that are predictive of the therapeutic outcome. Such predictive strategy is not available to decide whether anti-IgE (omalizumab) or anti-IL-5 (mepolizumab) should be prioritized in patients who are eligible to both therapies. In addition, the comparison of the magnitude of the clinical benefits achieved by these therapies remains unexplored in this population.

Study Design

The study is designed to initially randomly allocate patients from two strata (with or without maintenance oral corticosteroids) to oma- vs mepolizumab. According to the evaluation of response (at 4 or 6 months, respectively), subjects will then be either prolonged (for 12 months, for both therapies) on the same therapy, or switched to the other. For those who were switched, treatment will be prolonged (or not, in dual failers) after 4 or 6 months according to their evaluation of response. Time-points for analysis will be at 4 or 6 months, 10 months (interim analysis) and 18 or 22 months (final, posttreatment analysis).

State-of-the-art

Asthma is one of the most frequent chronic diseases, affecting 5 to 10% of the population worldwide. Omalizumab and mepolizumab represent the approved antibodies that are indicated in allergic and eosinophilic phenotypes of severe asthma respectively. However, if some patients fall into only one phenotypic category based on these criteria, a substantial number of patients are potentially eligible to both therapies. In those patients, no information is available to orientate towards a preferable therapy as the predictive weight of additional phenotypic traits, such as associated nasal polyps or early- versus late onset of disease, remains unknown. In addition, no head-to-head comparison of these therapies is available in this population.

Objectives of the study

Primary objectives To determine clinical features and blood (or sputum) biomarkers able to predict a better response to omalizumab or mepolizumab in severe asthma patients eligible to both therapies.

To determine the magnitude of response, in terms of improvement in symptoms, exacerbation rate and/or lung function, in responders to omalizumab vs mepolizumab.

Secondary objectives To compare the global baseline characteristics (clinical and biological features) of patients responding to omalizumab vs mepolizumab.

Management and reporting of adverse events.

If during the study, an adverse event (AE) (serious or non-serious) is identified as attributed to omalizumab or mepolizumab, this will be documented as appropriate in routine good clinical practice, to the Federal Agency of Medicines and Products of Health (AFMPS) as well as to the Central Ethic Committee.

Confidentiality of data.

The identity and participation of subjects will remain strictly confidential, according to Belgian laws dated 8 Dec 1992 related to the protection of private life and dated 22 Aug 2002 related to patient rights.

Specimens and associated data will be labeled with unique patient identification number.

Data will be anonymized in all files, results and publications related to the study.

The promoter confirms to authorize the regulatory surveillance, examination and controls by competent authorities, by allowing direct access to database/files, and this in full respect of confidentiality.

ELIGIBILITY:
Inclusion Criteria: • Signed informed consent form (ICF),

* Age >18+ years at time of signing ICF,
* Able to comply with the study protocol, in the investigator's judgment,
* Documented physician-diagnosed asthma ,
* Patients with severe disease and eligible to omalizumab and mepolizumab, and who have not yet received any of these therapies.

Exclusion Criteria:

* History of evidence of drug/substance abuse that would pose a risk to patient safety, interfere with the conduct of study, have an impact on the study results, or affect the patient's ability to participate in the study, in the opinion of the investigator
* Treatment with any investigational therapy within 6 months or 5 drug half-lives prior to enrolment.
* Known sensitivity to any of the active substances or their excipients to be administered during the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05-10 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy on asthma symptoms | Up to 22 months
  Asthma Control Test: 5 items of score 1 to 5 about symptoms, with result of 20 or above indicates good control; 15 to 19 indicates no good control and below 15 indicates no control at all, and a change of 3 points considered as clinically significant.
Efficacy on lung function | Up to 22 months
  Lung function measured as forced expiratory volume in one sec (FEV1), % predicted value (normal value of 80% predicted or above, and change of 100 mL considered as clinically significant).
Efficacy on severe exacerbations | Up to 22 months
  Number of exacerbation(s) per period of time (corrected per year) requiring systemic corticosteroid treatment for at least 3 days, and/or emergency visit or hospitalization for acute asthma.

SECONDARY OUTCOMES:
Predictive factors of therapeutic response | Baseline features (and according to response at 22 months)
  The putative predictive factors of therapeutic response to omalizumab or mepolizumab which will be assayed are the following: age at onset, year (> or < 30yrs); presence of nasal polyps, Y/N; blood eosinophils, n/microliter (< or > 300/microl); serum total IgE, units/L; serum periostin, ng/ml. A proteomic analysis will also be carried out on plasma samples.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Pilette, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (13):
- Belgium (13):
  - Universitair Ziekenhuis Brussel, Brussels, Brussels Capital
  - CHU de Charleroi, Charleroi, Hainaut
  - Grand Hôpital de Charleroi, Charleroi, Hainaut
  - Katholieke Universiteit Leuven, Leuven, Vlaams Brabant
  - AZ Delta Roeselare, Roeselare, West-vlaanderen
  - Centre Hospitalier Universitaire Saint Pierre, Brussels
  - Brugmann University Hospital, Brussels
  - Erasme University Hospital, Brussels
  - Cliniques universitaires St-Luc, Brussels
  - University Hospital, Ghent, Ghent
  - University Hospital of Liege, Liège
  - CHR Namur, Namur
  - Centre Hospitalier Universitaire Dinant Godinne - UCL Namur, Namur

IPD SHARING:
Plan to Share IPD: No